CLINICAL TRIAL: NCT02388386
Title: Pilot Study of Wireless Observed Therapy With an Ingestible Micro-Sensor Among Patients With Heart Failure and Left Ventricular Assist Devices
Brief Title: Monitoring Medication Adherence in Left Ventricular Assist Device Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Scripps Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROTEUS-LVAD
Record Dates: First submitted 2014-11-25; First posted 2015-03-17 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure; Medication Compliance
Keywords: Telemedicine; Mobile Health
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PROTEUS-SENSOR (Experimental): The current study is a prospective interventional design with a single experimental arm. The intervention consists of two components: an edible sensor and a wearable receiver health monitor.
  Interventions: Device: PROTEUS-SENSOR

INTERVENTIONS:
Device: PROTEUS-SENSOR — An edible sensor system, Proteus Digital™ has been developed for electronically confirming medication adherence, gathering physiologic metrics and communicating these data to patients. The system consists of two major components: an edible sensor and a wearable receiver health monitor. An electrical signal is activated upon ingestion of the Proteus Digital micro-sensor with transmission of this signal to a receiving abdominal patch to quantify medication compliance.

SUMMARY:
The investigators aim to develop a novel and wireless method for monitoring medication adherence among heart failure patients with left ventricular assist devices (LVADs). Proteus Digital™ has developed an ingestible and bio-absorbable micro-sensor as a strategy to monitor medication compliance. The edible sensor has at its core a silicon-based integrated circuit measuring 1.0 mm x 0.45 mm and is imbedded on a pill. Once ingested, this circuit is activated by gastric acid resulting in an electrochemical redox reaction and an electrical charge that is transmitted to a patch worn over the abdomen and wirelessly to a portable device such as a smart phone. This strategy of medication adherence differs from conventional adherence monitoring including pill counting and patient-recall by precisely tracking medication ingestion.

DETAILED DESCRIPTION:
The objectives are to assess the efficacy and safety of the Proteus Digital™ micro-sensor in an exploratory investigation among heart failure patients with LVADs. Medication adherence, specifically to anticoagulation is critically important in the post-implant period to maintain LVAD function and to decrease thromboembolic complications; however, commonly results in significant bleeding resulting in significant morbidity and mortality. In addition, the anticipated degree of anticoagulation is unpredictable after LVAD implantation due to factors related to changes in hepatic blood flow and endothelial dysfunction. Enrolling 10 patients will provide results into the function of micro-sensor and to provide a preliminary assessment of sensor-based activity, signal strength and signal duration in LVAD recipients. Participants will be enrolled during an in-patient hospitalization to assess the efficacy and safety of the device in a monitored setting.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing LVAD implantation for end-stage heart failure or admitted from the out-patient setting

Exclusion Criteria:

* Unable to consistently consume oral intake
* Hemodynamic instability defined as hypotension requiring intravenous vasoactive medications or arrhythmias requiring intravenous antiarrhythmics or oral antiarrhythmics for rhythm stabilization
* Gastrointestinal bleeding requiring intravenous gastric acid secretion inhibitors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Bhavnani, MD, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request

REFERENCES:
- [Background] Bhavnani SP, Narula J, Sengupta PP. Mobile technology and the digitization of healthcare. Eur Heart J. 2016 May 7;37(18):1428-38. doi: 10.1093/eurheartj/ehv770. Epub 2016 Feb 11. PMID 26873093
- [Background] DiCarlo LA, Weinstein RL, Morimoto CB, Savage GM, Moon GL, Au-Yeung K, Kim YA. Patient-Centered Home Care Using Digital Medicine and Telemetric Data for Hypertension: Feasibility and Acceptability of Objective Ambulatory Assessment. J Clin Hypertens (Greenwich). 2016 Sep;18(9):901-6. doi: 10.1111/jch.12787. Epub 2016 Feb 18. PMID 26890041
- [Background] DiCarlo L, Moon G, Intondi A, Duck R, Frank J, Hafazi H, Behzadi Y, Robertson T, Costello B, Savage G, Zdeblick M. A digital health solution for using and managing medications: wirelessly observed therapy. IEEE Pulse. 2012 Sep-Oct;3(5):23-6. doi: 10.1109/MPUL.2012.2205777. PMID 23014703
- [Background] Browne SH, Behzadi Y, Littlewort G. Let Visuals Tell the Story: Medication Adherence in Patients with Type II Diabetes Captured by a Novel Ingestion Sensor Platform. JMIR Mhealth Uhealth. 2015 Dec 31;3(4):e108. doi: 10.2196/mhealth.4292. PMID 26721413

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PROTEUS-SENSOR
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- PROTEUS-SENSOR: 10 consecutive heart failure patients with continuous flow left ventricular devices
Arm/Group | PROTEUS-SENSOR
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: System Performance - Positive Detection Accuracy
Description: Primary outcome measure of system performance will be estimated by the positive detection accuracy, defined as the number of ingestible sensors detected divided by those ingested
Time Frame: 30 minutes after ingestion
Measure: Number; unit: percentage of ingestions
Units Other Than Participants: Ingestions
Groups:
- Outcome Measure: Positive detection rate of 80%
Arm/Group | Outcome Measure
Number analyzed (Participants) | 10
Number analyzed (Ingestions) | 40
percentage of ingestions | 80

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Specific safety metrics will consist of the following composite outcome:
  1. Safety as measured by vital signs
  2. Cardiac rhythm monitoring review for arrhythmias
  3. LVAD device interrogation for changes in device parameters
  4. Implantable cardioverter defibrillator interrogation for arrhythmia occurrence
Time Frame: From time of ingestion to 30 minutes after ingestion
Population: Specific safety metrics will consist of the following composite outcome:
  1. Safety as measured by vital signs
  2. Cardiac rhythm monitoring review for arrhythmias
  3. LVAD device interrogation for changes in device parameters
  4. Implantable cardioverter defibrillator interrogation for arrhythmia occurrence
Measure: Count of Participants; unit: Participants
Groups:
- Vital Signs: Safety as measured by vital signs
- Cardiac Rhythm: Cardiac rhythm monitoring for arrhythmias
- LVAD Device Interrogation: Change in LVAD device parameters
- Implantable Cardioverter Defibrillator Interrogation: Assessment of cardiac arrhythmias by ICD interrogation
Arm/Group | Vital Signs | Cardiac Rhythm | LVAD Device Interrogation | Implantable Cardioverter Defibrillator Interrogation
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 hours
Description: Adverse events defined as nausea, abdominal pain after ingestion, skin irritation due to the adhesive patch, arrhythmia
Arm/Group | PROTEUS-SENSOR
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No